CLINICAL TRIAL: NCT05745597
Title: Prognostic Study of Different HPV Virus Integration in Women With HSIL
Brief Title: Prognostic Study of HPV Virus Integration in Women With HSIL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Maternity and Child Health Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HINH2301
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: HPV Infection; Virus Integration; HSIL, High Grade Squamous Intraepithelial Lesions
MeSH Terms: conditions — Papillomavirus Infections; Squamous Intraepithelial Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples from the cervix and vagina containing relevant cells, tissues and secretions, as well as peripheral blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HSIL (CIN2,3) women or cervical carcinoma in situ or early invasive carcinoma confirmed by pathology: In this study, women with pathologically confirmed HSIL(CIN2, 3) or women with cervical carcinoma in situ or early invasive cancer will be included. All participants will have four follow-up visits at enrollment and at months 6, 12, and 24.
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — Four samples of cervical exfoliated cells and fornix secretions were collected from all subjects at enrollment, 6 months, 12 months and 24 months for HPV integration status and vaginal microbiota diversity sequencing, and two additional samples of peripheral blood (whole blood + serum) were collected at enrollment.

SUMMARY:
Human papillomavirus (HPV) is currently one of the most common sexually transmitted infections, according to its carcinogenicity is divided into high-risk genotypes and low-risk genotypes, research has confirmed that carcinogenic HPV type continuous infection leads to a higher incidence of condyloma acuminatum and cervical cancer, while increasing the oropharyngeal cancer, vaginal cancer and other related cancer risk. Based on clinical practice, the purpose of this study was to: 1) identify the correlation between HPV integration and the outcome of disease in HSIL women. 2) To determine the prognostic value of different HPV gene integration status in HSIL women. 3) To clarify the relationship between different HPV gene integration status and diversity of vaginal flora in HSIL women.

DETAILED DESCRIPTION:
A total of 1000 women with HSIL were recruited from multiple centers. In this prospective cohort study, 4 samples of cervical exfoliated cells and fornix secretions were collected at enrollment, 6 months, 12 months and 24 months for HPV integration status and vaginal flora diversity sequencing, and 2 samples of peripheral blood (whole blood and serum) were collected at enrollment. The effects of HPV integration status and microbiota changes on the outcome and progression of HSIL were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed HSIL(CIN2, 3) in women or cervical carcinoma in situ or early invasive cancer;
* No surgical treatment or conization only;
* Obtain informed consent.

Exclusion Criteria:

* During pregnancy or lactation;
* Patients with a history of genital tract cancer;
* Previous history of hysterectomy, cervical surgery or pelvic radiotherapy;
* Received treatment related to genital tract infection, HPV or other STDs pathogen infection in the past one month;
* Use of antibiotics or vaginal microecological improvement products in the past 1 month.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pathologically confirmed HSIL(CIN2, 3) in women or cervical carcinoma in situ or early invasive carcinoma
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Cervical cytology testing at baseline | Baseline
  All participants were tested for cervical cytology at the time of baseline.
Cervical cytology testing at 6-month follow-up | 6-month follow-up
  All participants were tested for cervical cytology at 6-month follow-up for all participants.
Cervical cytology testing at 12-month follow-up | 12-month follow-up
  All participants were tested for cervical cytology at 12-month follow-up
Cervical cytology testing at 24-month follow-up | 24-month follow-up
  Cervical exfoliated cells and vaginal tissue samples were collected was performed at All participants were tested for cervical cytology at 24-month follow-up
16SrRNA sequencing of the vaginal secretions at baseline | Baseline
  All participants underwent vaginal secretion sequencing at baseline.
16SrRNA sequencing of the vaginal secretions at 6-month follow-up | 6-month follow-up
  All participants underwent vaginal secretion sequencing at 6-month follow-up
16SrRNA sequencing of the vaginal secretions at 12-month follow-up | 12-month follow-up
  All participants underwent vaginal secretion sequencing at 12-month follow-up
16SrRNA sequencing of the vaginal secretions at 24-month follow-up | 24-month follow-up
  All participants underwent vaginal secretion sequencing at 24-month follow-up
Human Papillomavirus (HPV) viral integration test at baseline | Baseline
  Human Papillomavirus (HPV) viral integration test was performed at baseline for all participants.
Human Papillomavirus (HPV) viral integration test at 6-month follow-up | 6-month follow-up
  Human Papillomavirus (HPV) viral integration test was performed at 6-month follow-up for all participants.
Human Papillomavirus (HPV) viral integration test at 12-month follow-up | 12-month follow-up
  Human Papillomavirus (HPV) viral integration test was performed at 12-month follow-up for all participants.
Human Papillomavirus (HPV) viral integration test at 24-month follow-up | 24-month follow-up
  Human Papillomavirus (HPV) viral integration test was performed at 24-month follow-up for all participants.
Human Papillomavirus (HPV) genotyping tests at baseline | Baseline
  All participants underwent Human Papillomavirus (HPV) genotyping tests at baseline.
Human Papillomavirus (HPV) genotyping tests at 6-month follow-up | 6-month follow-up
  All participants underwent Human Papillomavirus (HPV) genotyping tests at 6-month follow-up.
Human Papillomavirus (HPV) genotyping tests at 12-month follow-up | 12-month follow-up
  All participants underwent Human Papillomavirus (HPV) genotyping tests at 12-month follow-up.
Human Papillomavirus (HPV) genotyping tests at 24-month follow-up | 24-month follow-up
  All participants underwent Human Papillomavirus (HPV) genotyping tests at 24-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Pengming Sun, Study Chair — Fujian Maternal and Child Health Hospital
Locations (13):
- China (13):
  - Fujian Maternity and Child Health Hospital, Fuzhou, Fujian
  - Longyan First Hospital, Longyan, Fujian
  - Longyan People's Hospital, Longyan, Fujian
  - Nanping Second Hospital, Nanping, Fujian
  - Mindong Hospital of Ningde City, Ningde, Fujian
  - Ningde City Hospital, Ningde, Fujian
  - Affiliated Hospital of Putian University, Putian, Fujian
  - Putian First Hospital, Putian, Fujian
  - Sanming Second Hospital, Sanming, Fujian
  - Shenzhen Maternity and child Healthcare Hospital, Shenzhen, Guangdong
  - Shijiazhuang Obstetrics and Gynecology Hospital, Shijiazhuang, Hebei
  - Affiliated Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Maternal and Child Health Hospital of Hubei Province, Wuhan, Hubei